CLINICAL TRIAL: NCT04647630
Title: Prospective Study to Evaluate Streptococcus Pneumoniae Serotypes Prevalence in Community Acquired Pneumonia in Hong Kong Using a Urinary Kit
Brief Title: Evaluation of Streptococcus Pneumoniae Serotypes Prevalence Using a Urinary Kit
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Honoary Clinical Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2020.034
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAP: community acquired pneumonia
  Interventions: Diagnostic Test: urine test

INTERVENTIONS:
Diagnostic Test: urine test — test for pneumococcal antigen in urine

SUMMARY:
This is an epidemiology study for the prevalence and serotypes of pneumococcus pneumoniae in hospitalized patients with community acquired pneumonia (CAP). The serotypes of the pneumococcus pneumoniae will be determined by a urinary antigen assay. This is a single center, non-interventional observatory study.

DETAILED DESCRIPTION:
Patients admitted to the medical wards with a provisional diagnosis under "pneumonia","chest infection" or "fever" will be screened by research assistants.

Patients eligible with the inclusion criteria will be recruited into the study. Informed consent will be signed for those patients willing to participate in the study. Patient will be asked to save approximately 40 ml of urine. The urine sample will be processed in local laboratory and shipped out to a commercial lab for detection of any pneumococcal pneumoniae, and if present, serotyping will be performed at the same time using the same urine sample by urinary antigen assay. Meanwhile patients will be managed as usual by their clinical teams. Investigations and treatment will be offered by the clinical team as deemed necessary. The study team will only perform collection of urine and will not interfere the clinical management of the patients.

Positive results would be informed to the clinical teams for the appropriate action.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with signs and symptoms suggestive of pneumonia

Exclusion Criteria:

* 1. Nosocomial pneumonia which is acquired >= 48 hours after hospital admission. 2. Pneumonia which are already known to be caused by pathogens other than pneumococcus pneumoniae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults hospitalized with pneumococcal community acquired pneumonia (CAP)
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence of pneumococcal serotypes in adults hospitalized | 2 years
  Determine the prevalence of pneumococcal serotypes in adults hospitalized with pneumococcal community acquired pneumonia (CAP) using a specific urine antigen assay

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Shatin, Hong Kong